CLINICAL TRIAL: NCT04674852
Title: A Mayo-Designed Nonmetallic, Ultrasound-Detectable Marker for Metastatic Axillary Lymph Nodes in Breast Cancer
Brief Title: Mayo Designed Soft Tissue Ultrasound-Detectable Marker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christine U. Lee, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20-002505
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Breast Neoplasm Female; Ultrasound Therapy; Complications
Keywords: axillary lymph node; biopsy clip; biopsy marker; ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Marking cN+ nodes (Other): These patients have already undergone neoadjuvant chemotherapy for locally advanced breast cancer with metastasis to the axillary lymph nodes. During standard of care needle-directed I-125 seed localization, the research marker will also be deployed through the same needle. Ultrasound detection of the marker will be compared to conventional biopsy markers and the I-25 seed.
  Interventions: Device: Research Marker

INTERVENTIONS:
Device: Research Marker — The research marker is a cylindrical-shaped marker made of an FDA-approved material that can be seen by ultrasound.

SUMMARY:
Researchers are trying to determine if the Mayo marker is easily seen with ultrasound making it easier, faster, and more accurate for preoperative localization of the biopsied positive lymph node.

DETAILED DESCRIPTION:
Nonrandomized clinical trial to evaluate the Mayo-designed marker for ultrasound conspicuity at the time of preoperative ultrasound-guided localization.

Study participants are breast cancer patients with pathology-proven metastatic axillary lymph nodes. Per standard of care, a biopsy marker will have already been associated with the positive lymph node. 10 such patients scheduled for surgery at Mayo Clinic Rochester, MN with Dr. James Jakub will be enrolled. Preoperative radioactive seed localization will proceed as usual, but the marker will be additionally loaded with the seed into the needle using standard protocol. Before surgery, ultrasound will be performed to evaluate the marker.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older with breast cancer and biopsy-proven malignant involvement of an axillary lymph node
* Surgical management involves preoperative radioactive seed localization of a previously identified positive axillary lymph node
* Surgery will be performed by Dr. James Jakub at Mayo Clinic Rochester, MN
* Radioactive seed localization of an axillary lymph node.
* No contraception is necessary or required.
* English speaking

Exclusion Criteria:

* Scheduled for only radioactive seed localizations in the breast (as opposed to axilla)
* Are pregnant; although the twinkling marker is made of material widely used in orthopedic procedures, and hence, has an excellent safety profile, the investigators want to exclude the population of pregnant patients in this phase 0 clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Ultrasound detectability | Time of placement to surgical resection.
  Evaluation of ultrasound conspicuity of marker placed at time of radioactive seed localization.

SECONDARY OUTCOMES:
Conspicuity compared to conventional biopsy markers and radioactive seeds | Time of placement to surgical resection.
  To compare conspicuity of marker with that of conventional biopsy markers and I-125 localization seeds.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jakub JW, Hesley GK, Larson NB, Yaszemski MJ, Lee Miller A 2nd, Greenleaf JF, Urban MW, Lee CU. Ultrasonographic Detection and Surgical Retrieval of a Nonmetallic Twinkle Marker in Breast Cancer: Pilot Study. Radiol Imaging Cancer. 2022 Nov;4(6):e220053. doi: 10.1148/rycan.220053. PMID 36367449
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials